CLINICAL TRIAL: NCT07288645
Title: Enhancing Stability and Jumping Skills Through Combined Static and Dynamic Balance Training in Female Chinese University-Level Gymnastics Beginners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Wang (Other)
Responsible Party: Sponsor-Investigator, Yi Wang, Miss. Yi Wang, Principal Investigator, Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: USM/JEPeM/KK/25070591
Record Dates: First submitted 2025-11-15; First posted 2025-12-17 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Stability; Jumping Performance; Balance Training; Gymnastics Injury, Motor Learning, Balance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Static balance group (Experimental)
  Interventions: Behavioral: balance group
- Dynamic balance group (Experimental)
  Interventions: Behavioral: balance group
- Static and Dynamic balance group (Experimental)
  Interventions: Behavioral: balance group
- Control group (Active Comparator)
  Interventions: Behavioral: balance group

INTERVENTIONS:
Behavioral: balance group — An 8-week supervised training program conducted 2 times per week. Each 15-30 minute session comprises a combination of static balance exercises , dynamic balance exercises and Combining training. The intensity and difficulty of the exercises will be progressively increased throughout the intervention period.

SUMMARY:
This study aims to investigate the effects of different balance training programs (dynamic, static, combined dynamic and static) on the stability, jumping skills, and gymnastic movement skills of female university students who are beginners in gymnastics. Participants will be randomly divided into four groups: the first group will receive dynamic balance training (including exercises that maintain balance during movement); the second group will receive static balance training (including exercises that hold a fixed posture); the third group will receive combined dynamic and static balance training (including both static and dynamic balance exercises); and the fourth group will serve as a control group without additional balance training (or receive regular physical education classes as a control). The main outcomes to be measured before and after the training period are the participants' performance in specific stability tests, jumping tasks, and gymnastic movement skill assessments. The goal is to determine which balance training method (dynamic, static, or combined training) is most effective in improving the fundamental movement skills (including gymnastics-specific abilities) of gymnastics beginners.

ELIGIBILITY:
Inclusion Criteria:

1. Females
2. Age ranged between 18 -22 years old, normal body mass index (BMI) (18.5 -25kg/m²).
3. Undergraduate students of physical education at Beijing Sport University.
4. No prior systematic gymnastics training (or with ≤ 1 year of systematic training experience), and no history of congenital diseases or musculoskeletal injuries.

Exclusion Criteria:

1. Participants suffering from acute or chronic musculoskeletal injuries (lasting for 6 months or more), neurological disorders (such as epilepsy), or vestibular dysfunction.
2. Ranked athletes or elite athletes.
3. Participants with poor compliance (< 80%) who are unable to complete the 8 - week exercise intervention program.
4. Individuals who have recently undergone or are scheduled to undergo surgery within three months.

Ages: 18 Years to 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-11-06 (Actual); Primary Completion 2026-01-20 (Actual); Study Completion 2026-01-20 (Actual)

PRIMARY OUTCOMES:
The 8-point Star Offset (cm) | Baseline (pre-intervention) and at 8 weeks (immediately post-intervention)
Jump Height (cm) | Baseline (pre-intervention) and at 8 weeks (immediately post-intervention)
Peak Force (N) | Baseline (pre-intervention) and at 8 weeks (immediately post-intervention)
Rate of Force Development (N·S) | Baseline (pre-intervention) and at 8 weeks (immediately post-intervention)
Impulse (N·s) | Baseline (pre-intervention) and at 8 weeks (immediately post-intervention)

SECONDARY OUTCOMES:
Center of gravity deviation distance (mm) | Baseline (pre-intervention) and at 8 weeks (immediately post-intervention)
Joint Angle variation (°) | Baseline (pre-intervention) and at 8 weeks (immediately post-intervention)
Vertical Jump Efficiency (%) | Baseline (pre-intervention) and at 8 weeks (immediately post-intervention)
Landing Impact Force (N) | Baseline (pre-intervention) and at 8 weeks (immediately post-intervention)
Body Oscillation Amplitude (mm) | Baseline (pre-intervention) and at 8 weeks (immediately post-intervention)
Rotation Smoothness Index (°) | Baseline (pre-intervention) and at 8 weeks (immediately post-intervention)
Height (cm) | Baseline (pre-intervention) and at 8 weeks (immediately post-intervention)
Weight (kg) | Baseline (pre-intervention) and at 8 weeks (immediately post-intervention)
BMI (kg/m2) | Baseline (pre-intervention) and at 8 weeks (immediately post-intervention)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Sport University, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Related Info — https://ejepem.usm.my/myapplication

DOCUMENTS (2):
  • Study Protocol (2025-09-25): https://cdn.clinicaltrials.gov/large-docs/45/NCT07288645/Prot_000.pdf
  • Informed Consent Form (2025-11-06): https://cdn.clinicaltrials.gov/large-docs/45/NCT07288645/ICF_001.pdf